CLINICAL TRIAL: NCT01815047
Title: Vitamin D Status Impacts Inflammation and Risk of Infections During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB 1201002753; USDA 2012-67017-30216 (Other Grant/Funding Number: USDA 2012-67017-30216)
Record Dates: First submitted 2013-03-11; First posted 2013-03-20 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Inflammation; Infection
Keywords: Vitamin D; Pregnancy; Inflammation; Infection; Placenta; Cytokine; Microbiome
MeSH Terms: conditions — Inflammation; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 200 IU Vitamin D3 (Experimental): A singular daily dose of 200 IU vitamin D3
  Interventions: Dietary Supplement: Vitamin D3 Supplementation
- 2000 IU Vitamin D3 (Experimental): A singular daily dose of 2000 IU vitamin D3
  Interventions: Dietary Supplement: Vitamin D3 Supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D3 Supplementation

SUMMARY:
The goal of this study is to characterize the function and efficacy of the bioactive nutrient, vitamin D, in relation to infection and inflammatory status across pregnancy. The three specific aims of this study are 1) To address the impact of maternal vitamin D status on inflammation and infections across pregnancy using retrospective data, 2) To address the impact of vitamin D supplementation on maternal vitamin D status, inflammation and infections across pregnancy using prospective data and 3) To assess the impact of maternal vitamin D status during pregnancy on inflammatory mediators at the level of the placenta.

DETAILED DESCRIPTION:
Archived serum collected from 158 adolescents at mid-gestation (approximately 26 weeks) and delivery will be analyzed for inflammatory cytokines. The impact of these inflammatory markers will be assessed by comparing the data to measures of vitamin D (25(OH)D, calcitriol and parathyroid hormone) and infections and inflammatory complications abstracted from medical charts. Placental samples were collected from a subset (n=132) of these pregnant teens and these tissues will be analyzed using genome wide microarray of messenger ribonucleic acid (mRNA) and microRNA (miRNA) related to inflammatory processes. A separate group of pregnant adolescents (n=140) will be recruited at entry into prenatal care for a vitamin D supplementation trial. Teens will be randomly assigned to one of two supplements (200 IU D3/d vs. 2000 IU D3/d). Similar to the retrospective analysis, maternal calciotropic hormones and inflammatory cytokines will be assessed at entry into the study, mid-gestation (23-28 weeks) and at delivery. Inflammatory processes and infections reported across pregnancy will be evaluated in relation to vitamin D status and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents between 13 and 18 years of age
* Between 12 and < 30 weeks pregnant

Exclusion Criteria:

* HIV-infection
* Eating disorders
* Malabsorption diseases
* Diabetes mellitus
* Gestational diabetes
* Pregnancy induced hypertension or elevated diastolic blood pressure (>110)
* Steroid use
* Substance abuse history
* Taking medications known to influence Ca or vitamin D status
* Diagnosis of elevated blood lead concentrations during childhood
* Smokes tobacco

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in Vitamin D status, infections and inflammation across pregnancy after Vitamin D supplementation | Entry into study, mid-gestation and delivery
  Maternal calciotropic hormones (25(OH)D, 1,25(OH)2D, 24,25(OH)2D, and PTH) and inflammatory cytokines (CRP, interleukin [IL]-6 and IL-10 and tumor necrosis factor [TNF]-alpha) will be measured at entry into the study and again at 23-28 weeks gestation and delivery after treatment with 200 IU or 2000 IU D3/d. These measures will be compared to inflammatory processes and infections reported in medical records across pregnancy.

SECONDARY OUTCOMES:
Change in maternal vitamin D status and inflammatory markers in serum | Mid-gestation and delivery
  In a retrospective analysis, inflammatory cytokines (CRP, IL- 6 and IL-10 and TNF-alpha) in archived serum collected from a cohort of 158 adolescents that were longitudinally followed across pregnancy both at mid-gestation and at delivery will be related to 25-hydroxyvitamin D (25(OH)D), 1,25- dihydroxyvitamin D (1,25(OH)2D) and parathyroid hormone (PTH) and medically treated infections and inflammatory conditions abstracted from medical records.
Association of maternal vitamin D status (25(OH)D concentration with longitudinal change in 1,25(OH)2D, PTH, 24,25(OH)2D,and the vitamin D metabolite ratio | Mid-gestation and delivery

OTHER OUTCOMES:
Vitamin D and placental inflammation | Delivery
  Genome-wide microarray studies of mRNA and miRNA in a subset of placental tissue from adolescents with insufficient (<15 ng/mL) and sufficient vitamin D status (>30 ng/mL) will be screened for differential regulation of genes and gene networks involved in inflammatory processes.
Vaginal microbiome profile | Mid to late gestation
  Vitamin D supplementation (200 IU/d D3 and 2000 IU/d D3), dietary intake, 25-hydroxyvitamin D (25(OH)D), 1,25-dihydroxyvitamin D (1,25 (OH)2D), parathyroid hormone(PTH), inflammatory cytokines (CRP, IL- 6 and IL-10 and TNF-alpha) and infection (from medical records) will be related to vaginal microbiome profile.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O'Brien, PhD, Principal Investigator — Cornell University
Locations (1):
- Highland Hospital, Rochester, New York, United States

REFERENCES:
- [Derived] Best CM, Pressman EK, Queenan RA, Cooper E, Vermeylen F, O'Brien KO. Gestational Age and Maternal Serum 25-hydroxyvitamin D Concentration Interact to Affect the 24,25-dihydroxyvitamin D Concentration in Pregnant Adolescents. J Nutr. 2018 Jun 1;148(6):868-875. doi: 10.1093/jn/nxy043. PMID 29796622